CLINICAL TRIAL: NCT05973110
Title: Examining the Efficacy of a Virtual Reality Cognitive Remediation Program for People Living With Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); The Royal's Institute of Mental Health Research (Other)
Responsible Party: Principal Investigator, Synthia Guimond, Scientist, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023001
Record Dates: First submitted 2023-07-04; First posted 2023-08-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Psychotic Disorders; Schizophrenia; Schizo Affective Disorder
Keywords: Psychotic Disorders; Cognitive Remediation; Virtual Reality; Neurocognition; Social Cognition; Community Functioning
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either 12 sessions over 6 weeks of a cognitive remediation intervention or 12 sessions over 6 weeks of an active control intervention. Both conditions will involve activities in virtual reality.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the clinical trial, the study staff members delivering the intervention are unable to remain blind and are the only individuals who will be aware of the study arm assignment. Assessment staff members, investigators, and participants will be blinded to study arm assignment and will never be involved in the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Remediation (Experimental)
  Interventions: Behavioral: Cognitive Remediation
- Active Control (Active Comparator)
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Cognitive Remediation — In each of the 12 visits, participants will complete exercises in virtual reality for two sessions of about 15 minutes separated by a break of 5 to 10 minutes. Participants then engage in a bridging conversation with study staff for about 15 minutes. More details about each condition will be added after study completion to protect the blinding of our participants.
  Arms: Cognitive Remediation
Behavioral: Active Control — In each of the 12 visits, participants will complete exercises in virtual reality will complete exercises in virtual reality for two sessions of about 15 minutes separated by a break of 5 to 10 minutes. Participants then engage in a bridging conversation with study staff for around 10 to 15 minutes. More details about each condition will be added after study completion to protect the blinding of our participants.
  Arms: Active Control

SUMMARY:
Individuals living with a psychotic disorder often experience changes to their thinking and social skills that can lead to challenges with work, school, relationships and living independently. One intervention to target these areas is cognitive remediation therapy, which can be delivered in virtual reality to help apply the skills and strategies learned to day-to-day life. Over the past few years, our team has co-developed a cognitive remediation program in virtual reality with healthcare professionals and people with lived experiences of psychosis. The current trial tests the feasibility and efficacy of this cognitive remediation program in virtual reality at improving thinking skills, social skills, and daily life functioning.

DETAILED DESCRIPTION:
Eligible participants will be administered various clinical (including a module from the Mini International Neuropsychiatric Interview and the Wechsler Abbreviated Scale Intelligence (WASI) to confirm eligibility), neurocognitive, social-cognitive, and community functioning assessments across two baseline visits. Participants are then randomly assigned to one of two study arms (a cognitive remediation intervention and active control, both using virtual reality). Regardless of the study arm assignment, participants will complete a six weeks (12 visits) training program where they will complete exercises in virtual reality and converse with study staff about a pre-selected topic. After each training visits, participants will also complete short questionnaires about their experience. One-week and three-months post-intervention, participants will complete the same assessments administered during the baseline visits. Also, at the one-week post-intervention time point, participants will complete a satisfaction with cognitive remediation program questionnaire.

The investigators will also use ecological momentary assessments (EMAs) delivered through a smartphone app to measure changes in thinking skills and daily life functioning within the context of this clinical trial. At the first visit, the investigators will invite participants to download the EMA app, DigiSensing, to their phone. DigiSensing is built from the open access MindLamp app, which has been used to measure neurocognition in previous studies. Through the DigiSensing app, the investigators will deliver three, ten-minute assessments at baseline, one-week post-intervention, and six-months post-intervention. Each assessment has thinking skill tasks, and questions about mood, clinical symptoms, thinking skills, and daily life functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a psychosis-spectrum disorder
* Equal or between 20 to 55 years old
* Ability to read and speak English
* Be clinically stable, as defined as a total Positive And Negative Severity Symptoms score equal or between 30 - 95
* No changes to their medication dosage, starting a new medication, or stopping a medication within the past month before signing the consent form

Exclusion Criteria:

* Neurological or medical disorders that may produce cognitive impairment
* Intellectual disability or a score equal or below 70 on the Wechsler Abbreviated Scale of Intelligence.
* Any vision conditions that cannot be corrected with contact lenses or glasses that can fit in the virtual reality googles.
* Past history of seizures, fit, and epilepsy
* Any severe medical condition related to the eyes, ears, and balance
* History of substance use disorder within the last 3 months
* Past traumatic brain injury resulting in a loss of consciousness
* Do not own a smartphone

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in neurocognitive performance from baseline to 1-week and 3-months post- intervention (Cambridge Automated Neuropsychology Battery). | Participants complete the Cambridge Automated Neuropsychology Battery at baseline, 1-week post-intervention, and 3-months post-intervention
  The investigators will measure neurocognition using nine subtests from the Cambridge Automated Neuropsychology Battery, in which a composite z-score will be computed to represent the cognitive domains measured.
Change in social-cognitive performance from baseline to 1-week and 3-months post-intervention (PENN emotion recognition task). | Time Frame: Participants complete the PENN emotion recognition task at baseline, 1-week post-intervention, and 3-months post-intervention
  The investigators will measure the social cognition domain, emotion recognition, using the PENN emotion recognition task. The total score ranges from 0 to 40, with higher scores indicating greater emotion recognition ability.
Change in social cognition performance from baseline to 1-week and 3-months post-intervention (Ambiguous Intentions Hostility Questionnaire). | Participants complete the Ambiguous Intentions Hostility Questionnaire at baseline, 1-week post-intervention, and 3-months post-intervention
  The investigators will measure the social cognition domain, attribution bias, using the Ambiguous Intentions Hostility Questionnaire. The Ambiguous Intentions Hostility Questionnaire is rated on a Likert Scale. The total score ranges from 3 to 16, with higher scores indicating greater blame, perceived intention, and anger.
Change in social cognition performance from baseline to 1-week and 3-months post-intervention (Emotion Regulation Questionnaire). | Participants complete the Emotion Regulation Questionnaire test at baseline, 1-week post-intervention, and 3-months post-intervention.
  The investigators will measure the social cognition domain, emotion regulation, using the Emotion Regulation Questionnaire. Each of the 10 items of the Emotion Recognition Questionnaire is rated on a 7-point Likert scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The total score ranges from 10 to 70, with higher scores indicating a greater emotion regulation abilities.
Change in social cognition performance from baseline to 1-week and 3-months post-intervention (The Hinting Task). | Participants complete the Hinting Task test at baseline, 1-week post-intervention, and 3 months post-intervention
  The investigators will measure the social cognition domain, theory of mind, using the The Hinting Task. Each of the 10 items of the Hinting Task is scored on a scale from 0 to 2. The total score ranges from 0 to 20 with higher scores indicating greater theory of mind abilities.
Change in the community functioning performance from baseline to 1-week and 3-months post-intervention (UCSD performance-based skills assessment brief). | Participants complete the measure at baseline, 1-week post-intervention, and 3 months post-intervention.]
  The investigators will measure community functioning through the UCSD performance-based skills assessment brief. The total score is from 0 to 100 with higher score indicating a greater performance in community functioning.
Change in the community functioning performance from baseline to 1-week and 3-months post-intervention ( modified Global Assessment of Functioning Scale). | Participants complete the modified Global Assessment of Functioning at baseline, 1-week post-intervention, and 3-months post-intervention
  The investigators will measure community functioning through the modified Global Assessment of Functioning Scale. The total score is from 0 to 100 with higher score indicating a greater functioning.
Change in the community functioning performance from baseline to 1-week and 3-months post-intervention (Role Functioning Scale). | Participants complete the Role Functioning Scale at baseline, 1-week post-intervention, and 3-months post-intervention.
  The investigators will measure community functioning through the Role Functioning Scale. Each of the 4 items of the Role Functioning Scale is scored on a scale of 1 to 7. The total score is from 4 to 28 with a higher score indicating a greater community functioning.
Feasibility of the Intervention (attrition rate). | The training completion will be computed at the 1-week post-intervention timepoint.
  The investigators will measure the feasibility of the intervention by verifying adherence and attrition of participants. The percentage of participants who completed the training program will be computed after the participant completes their final intervention visits.
Feasibility of the intervention (homework completion). | Homework completion will be computed at the 1-week post-intervention timepoint.
  The investigators will measure the feasibility of the intervention by verifying the homework completion by participants. The percentage of homework completion will be computed after the participant completes their final intervention visit.
Feasibility of the intervention (cybersickness). | Participants complete the Simulator Sickness Questionnaire at each intervention visit, which is scheduled twice a week for six weeks. The composite mean score will be computed at the 1-week post-training time point for each participant.
  The investigators will measure the feasibility of the intervention by creating a composite mean score of cybersickness reported on the Simulator Sickness Questionnaire for each participant. The Simulator Sickness Questionnaire is composed of 16, four-point Likert scale items with responses ranging from "never" to "severe". A higher score on the Simulator Sickness Questionnaire indicates greater cybersickness experienced.
Acceptability of the intervention | The satisfaction questionnaire will be administered at the 1-week post-intervention time point.
  The acceptability of the intervention will be measured through a study-specific satisfaction with cognitive remediation intervention questionnaire.
Change in the acceptability of the intervention from the sixth intervention visit (3 weeks in intervention) to 1-week post-intervention. | The Treatment Acceptability/Adherence Scale will be administered at the sixth intervention visit (3 weeks in the intervention) and 1-week post-intervention.
  The acceptability of the intervention will be measured through the Treatment Acceptability/Adherence Scale (TAAS). Each of the 10 items of The Treatment Acceptability/Adherence Scale is rated on a 7-point Likert-type scale, with responses ranging from 1 ("strongly disagree") to 7 ("strongly agree "). The total score ranges from 10 to 70 with higher score indicating greater acceptability of treatment and greater anticipated ability to adhere to it.

SECONDARY OUTCOMES:
Feasibility of Integrating EMAs into a Clinical Trial | The completion of the EMA surveys will be computed at the 6-months post-intervention timepoint.
  The investigators will assess the feasibility of integrating EMAs into a clinical trial by calculating the overall completion rate of the EMA survey (number of EMA surveys completed divided by the total number of EMA surveys).
Change in the EMA Neurocognition performance from baseline to 1-week and 6-months post-intervention - Jewel task | Participants complete the Jewels task through the DigiSensing App at baseline, 1-week post-intervention, and 6-months post-intervention.
  The investigators will measure neurocognition through the EMA survey using a Jewels Trail test, which is modelled after the Trail Making Test. A greater response time on the Jewels Trail test indicates decreased neurocognitive performance.
Change in the EMA Community Functioning performance from baseline to 1-week and 6-months post-intervention ( Questionnaire about Process to Recovery). | Participants complete the Questionnaire about Process to Recovery through the DigiSensing app at baseline, 1-week post-intervention, and 6-months post-intervention
  The investigators will measure community functioning through the EMA survey using the Questionnaire about Process to Recovery. Each of the 15 items of the Questionnaire about Process to Recovery is rated on a 4-point Likert-type scale, with responses ranging from 0 ("disagree strongly") to 4 ("agree strongly"). The total score ranges from 0 to 60, with higher scores indicating a greater recovery.
Change in the EMA Community Functioning performance from baseline to 1-week and 6-months post-intervention (Social Functioning Questionnaire). | Participants complete the Social Functioning Questionnaire through the DigiSensing app at baseline, 1-week post-intervention, and 6-months post-intervention.
  The investigators will measure community functioning through the EMA survey using the Social Functioning Questionnaire.Each of the 8 items of the Social Functioning Questionnaire is scored on a scale ranging from 0 to 3 points. The total score ranges from 0 to 24 with higher scores representing poorer social functioning.

OTHER OUTCOMES:
Symptom Severity at baseline | Participants complete the Positive and Negative Severity Scale at baseline.
  The investigators will measure symptom severity through the Positive and Negative Severity Scale. Each of the 30 items of the Positive and Negative Severity Scale is rated on a scale of 7 points and the total score ranges from 30 to 210, with higher scores indicating more severe psychotic disorder symptoms.
Change in Symptom Severity from baseline to 1-week post-intervention and 3-months post-intervention. | Participants complete the brief version of the Positive and Negative Severity Scale at 1-week post-intervention and 3-months post-intervention.
  The investigators will measure symptom severity through the brief version of the PANSS (PANSS-6). Each of the 6 items of the brief version of the Positive and Negative Severity Scale is rated on a scale of 7 points and the total score ranges from 6 to 42 with higher scores indicating more severe symptoms of a psychotic disorder.
Change in Self-Reported Neurocognition performance from baseline to 1-week, 3-months and 6-months post intervention- Subjective Scale to Investigate Cognition in Schizophrenia - Brief. | Participants complete the Subjective Scale to Investigate Cognition in Schizophrenia - Brief at baseline, 1-week post-intervention, 3-months post-intervention, and 6-months post-intervention.
  The investigators will measure subjective perceptions of neurocognitive functioning through the Subjective Scale to Investigate Cognition in Schizophrenia - Brief (SSTICS-Brief). Each of the 14 items are scored on a 5 points Likert-type scale that extends from 0 ("never") to 4 ("very often"). The total score ranges from 0 to 56 with higher score indicating a higher perceived difficulty in neurocognition.
Intrinsic Motivation | Participants complete the Intrinsic Motivation Inventory for Schizophrenia Research at baseline.]
  The investigators will measure motivation through the Intrinsic Motivation Inventory for Schizophrenia Research (IMI-SR). The Intrinsic Motivation Inventory for Schizophrenia Research (IMI-SR) is rated on a 7-point Likert-type scale with responses ranging from 1 ("not at all true") to 7 ("very true"). The score ranges from 30 to 210 with higher scores indicating greater intrinsic motivation.
Motivation | Participants complete the Basic Psychological Need Satisfaction and Frustration Scale at baseline.]
  The investigators will measure motivation through the Basic Psychological Need Satisfaction and Frustration Scale. Each item is scored on a 5 points Likert-type scale that extends from 1 ("Not true at all") to 5 ("Completely true"). An overall composite score will be created, with scores ranging from 1 to 6. Higher scores indicate greater satisfaction of the psychological needs for autonomy, competence, and relatedness.
Social Support (Friends) | Participants complete the Perceived Social Support from Friends at baseline.
  The investigators will measure perceived social support through the Perceived Social Support from Friends scale. Each of the 20 items has a maximum score of 1 ("yes", "no", and "don't know" response items). The scores range from 0 to 20 with higher scores indicating greater perceived social support from friends.
Social Support (Family) | Participants complete the Perceived Social Support from Family at baseline.
  The investigators will measure perceived social support through the Perceived Social Support from Family scale. Each of the 20 items has a maximum score of 1 ("yes", "no", and "don't know" response items). The scores range from 0 to 20 with higher scores indicating greater perceived social support from family.
Change in level of stress performance from baseline to 1-week and 3-months post-intervention (Perceived Stress Scale). | Participants complete the Perceived Stress Scale at baseline, 1-week post-intervention, and 3-months post-intervention.
  The investigators will measure the level of stress through the Perceived Stress Scale. The Perceived Stress Scale is rated on a five-point scale from 0 ("never") to 4 ("very often"). Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Change in stress resilience performance from baseline to 1-week and 3-months post-intervention (Brief Resilience Scale). | Participants complete the Brief Resilience Scale at baseline, 1-week post-intervention, and 3-months post-intervention.
  The investigators will measure stress resilience through the Brief Resilience Scale. The Brief Resilience Scale is rated on a scale from 1 ("low resilience") to 5 ("high resilience"). The total mean score ranges from 1 to 5 with a higher score indicating a higher resilience.
Affect | Participants complete the Core Affect Grid at each intervention visit, which is scheduled twice a week for six weeks. The composite mean score will be computed at the 1-week post-training time point for each participant
  The investigators will measure the level of affect arousal by creating a composite mean score reported on a core affect grid for each participant. The Core Affect Grid is composed with two dimensions measuring the level of arousal and pleasantness and is rated on a 5 points scale. A higher score indicates greater pleasure or arousal.
Change in the Therapeutic Alliance from sixth intervention (3-weeks in the intervention) to 1-week post-intervention | Participants complete the Work Alliance Inventory Short version at the sixth intervention visit (3 weeks in the intervention) and 1-week post-intervention.
  The investigators will measure the therapeutic alliance through the Work Alliance Inventory (WAI-S). The Work Alliance Inventory is rated on a 7-point Likert-type scale with responses ranging from 0 ("never") to 7 ("always"). The total score is from 7 to 84 with higher score indicating a greater work alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Synthia Guimond, PhD, Principal Investigator — Royal Ottawa Mental Health Centre
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected from this study may be shared with other researchers at the Royal's Institute of Mental Health Research for analyses and re-analyses. Variables of the study and scripts used for analyses will be made available to the public. De-identified data will also be shared with the general public and researchers upon request. Data that can connect with participants' identity will NOT be used or shared for analyses.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will become available upon completion of the study and once results have been published in an academic journal (anticipated year of publication: 2026).
Access Criteria: Upon request to Synthia Guimond

REFERENCES:
- [Background] Jahn FS, Skovbye M, Obenhausen K, Jespersen AE, Miskowiak KW. Cognitive training with fully immersive virtual reality in patients with neurological and psychiatric disorders: A systematic review of randomized controlled trials. Psychiatry Res. 2021 Jun;300:113928. doi: 10.1016/j.psychres.2021.113928. Epub 2021 Apr 6. PMID 33857847
- [Background] National Institute of Mental Health (n.d.). Schizophrenia. https://www.nimh.nih.gov/health/topics/schizophrenia
- [Background] Viertio S, Tuulio-Henriksson A, Perala J, Saarni SI, Koskinen S, Sihvonen M, Lonnqvist J, Suvisaari J. Activities of daily living, social functioning and their determinants in persons with psychotic disorder. Eur Psychiatry. 2012 Aug;27(6):409-15. doi: 10.1016/j.eurpsy.2010.12.005. Epub 2011 Mar 5. PMID 21377336
- [Background] Schroeder AH, Bogie BJM, Rahman TT, Therond A, Matheson H, Guimond S. Feasibility and Efficacy of Virtual Reality Interventions to Improve Psychosocial Functioning in Psychosis: Systematic Review. JMIR Ment Health. 2022 Feb 18;9(2):e28502. doi: 10.2196/28502. PMID 35179501
- [Background] Shvetz C, Gu F, Drodge J, Torous J, Guimond S. Validation of an ecological momentary assessment to measure processing speed and executive function in schizophrenia. NPJ Schizophr. 2021 Dec 21;7(1):64. doi: 10.1038/s41537-021-00194-9. PMID 34934063
- [Background] Torous, J., Wisniewski, H., Bird, B., Carpenter, E., David, G., Elejalde, E., Fulford, D., Guimond, S., Hays, R., Henson, P., Hoffman, L., Lim, C., Menon, M., Noel, V., Pearson, J., Peterson, R., Susheela, A., Troy, H., Vaidyam, A., & Weizenbaum, E. (2019). Creating a Digital Health Smartphone App and Digital Phenotyping Platform for Mental Health and Diverse Healthcare Needs: an Interdisciplinary and Collaborative Approach. Journal of Technology in Behavioral Science, 4(2), 73-85. https://doi.org/10.1007/s41347-019-00095-w
- [Background] Yee, J., Matheson, H., Bogie, B. J. M., Thérond, A., Charest, M., van Driel, C., Lei, Y-T., Noël, C., Goyette, M., Cretu, A. M., Tremblay, S., Morris, C., Attwood, D., Baines, A., Stewart, A., Bouchard, S., Bowie, C.R., & Guimond, S. (2023). The development of a user-centered and co-designed virtual reality cognitive remediation program for people living with a psychotic disorder [Manuscript in preparation]. Institute of Mental Health Research, The Royal Ottawa Mental Health Centre.